CLINICAL TRIAL: NCT06788704
Title: The Effect of Tadalafil 5 mg on Erection and Persistent Storage Lower Urinary Tract Symptoms After Transurethral Resection of Prostate: a Randmized Controlled Trial
Brief Title: Tadalafil Daily Used Post Turp
Status: Completed | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelhalim Elsayed, assistant lecturer of urology, Kafrelsheikh University
Other Study IDs: Tadalafil daily used post turp
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Erectile Dysfunction Following Urethral Surgery
MeSH Terms: interventions — Tadalafil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient recive tadalafil 5mg once daily early post turp
  Interventions: Drug: Tadalafil 5mg
- Patient recive placebo once daily early post turp
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil 5mg — Patient recive tadalafil 5mg once daily early post turp
  Groups: Patient recive tadalafil 5mg once daily early post turp
Drug: Placebo — Patient recive placebo once daily early post turp
  Groups: Patient recive placebo once daily early post turp

SUMMARY:
to assess the effect of early tadalafil 5 mg once daily on persistent storage lower urinary tract symptoms (LUTS) and erectile function after transurethral resection of the prostate (TURP).

ELIGIBILITY:
Inclusion Criteria:

* sexual active men

Exclusion Criteria:

* sexual inactive men
* cardiac patients

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: Sexual active male patients underwent TURP
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Assess erectile function | One month
  Using IIEF score
Assess erectile function | 3 month
  Usine IIEF score

SECONDARY OUTCOMES:
Assess storage symptoms | One month
  Using IPSS Score
Assess storage symptoms | 3 month
  Using IPSS score

CONTACTS AND LOCATIONS:
Locations (1):
- Elsayed Abdelhalim Elsayed, Zagazig, Egypt

REFERENCES:
- [Derived] Taha DE, Nabeeh H, Zeinelabden KM, Abdelhalim E, Elmekawy S, Samaha II, Behiry A, Elmoaty AA, Abdelbaky T, Ibrahim A. The effect of tadalafil 5 mg on erection and persistent storage lower urinary tract symptoms after transurethral resection of prostate: a randomized controlled study. Basic Clin Androl. 2025 Jul 1;35(1):27. doi: 10.1186/s12610-025-00273-2. PMID 40588736